CLINICAL TRIAL: NCT06670586
Title: Assessment of Reproductive and Perinatal Outcomes According to the Fertilisation Technique in Non-Male Factor Infertility Patients: Conventional in Vitro Fertilisation Versus Intracytoplasmic Sperm Injection
Brief Title: Assessment of Reproductive Outcomes in Non-Male Factor Infertility Patients: Conventional in Vitro Fertilisation Versus Intracytoplasmic Sperm Injection
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Dolores Cuquerella Fernandez-Vazquez (Other)
Responsible Party: Sponsor-Investigator, Maria Dolores Cuquerella Fernandez-Vazquez, Principal Investigator, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21/707-E
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: In Vitro Fertilization; Infertility Assisted Reproductive Technology
Keywords: In Vitro Fertilization; ICSI; randomized controlled trial; sibling oocytes
MeSH Terms: interventions — Congresses as Topic; Fertilization in Vitro; Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Intervention Model Description: Oocytes obtained from every participant are divided in two groups and each group is randomly allocated to one of the two techniques that we want to analyze. So, there are not two groups of participants but two groups of oocytes from every participan
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional IVF (cIVF) (Active Comparator): The oocytes of this arm will be fertilized using conventional In Vitro Fertilization (cIVF)
  Interventions: Procedure: conventional in vitro fertilization
- Intracytoplasmic Sperm Injection (ICSI) (Active Comparator): The oocytes of this arm will be fertilized using Intracytoplasmic Sperm Injection (ICSI)
  Interventions: Procedure: intracytoplasmic sperm injection (ICSI)

INTERVENTIONS:
Procedure: conventional in vitro fertilization — Fertilization via conventional In Vitro Fertilization
  Arms: conventional IVF (cIVF)
Procedure: intracytoplasmic sperm injection (ICSI) — Fertilization via intracytoplasmic sperm injection
  Arms: Intracytoplasmic Sperm Injection (ICSI)

SUMMARY:
The aim of this clinical trial is to evaluate the efficiency of two fertilization techniques used in Assisted Reproduction: conventional In Vitro fertilization (cIVF) and Intracytoplasmic Sperm Injection (ICSI), in terms of in-vitro and clinical results, in non-male infertility patients, comparing them in sibling oocytes.

The main questions it aims to answer are:

Does ICSI result in better fertilization rate, blastocyst rate or usable blastocyst rate? Does ICSI result in better pregnancy, clinical pregnancy and live birth rates?

Researchers will compare cIVF to ICSI in sibling oocytes to assess if a technique offers better results.

Participants undergoing an IVF/ICSI cycle will have their oocytes randomly divided in two groups: the oocytes from one group will be fertilized using cIVF and the oocytes from the other group using ICSI.

DETAILED DESCRIPTION:
It is a prospective randomized study performed in the Reproduction Unit of Hospital Clinico San Carlos, in Madrid.

The study involves In Vitro Fertilization cycles with at least 6 oocytes retrieved and with normal semen parameters according to WHO.

The objective is to compare conventional In Vitro Fertilization (cIVF) and Intracytoplasmic Sperm Injection (ICSI) in sibling oocytes from the same cohort.

The oocytes obtained after the ovum pick up will be randomly divided in two groups and the fertilization technique (cIVF or ICSI) will be randomly assigned to each group.

Maturity stage, fertilization and embryo development to blastocyst will be individually recorded for every oocyte. Additionally, the destination of every embryo (transferred, cryopreserved or discarded) will be registered. This decision will be based just on embryo quality, irrespective of the fertilization technique.

MII rate, blastocyst rate and usable blastocyst (transferred or cryopreserved) rate will be calculated for each group.

Additionally, embryo transfers will be performed in the fresh cycle or in the associated thaw cycles using the cryopreserved embryos. In every transfer, the technique used to obtain the transferred embryo will be registered.

The results of the embryo transfers will be recorded as pregnancy (positive beta-hCG 14 days after transfer), clinical pregnancy (diagnosed by ultrasonographic visualization of a gestational sac 4 weeks after transfer, including ectopic pregnancy) and live birth delivery (deliveries with at least one live birth). Pregnancy rate, clinical pregnancy rate and live birth delivery rate will be calculated for each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 6 fresh, own oocytes.
* Patients with culture to blastocyst stage for all the embryos.
* Non-male factor infertility patients: semen sample with a good progresive sperm count, appropriate for cIVF.

Exclusion Criteria:

* Patients not willing to sign the informed consent. Patients not understanding Spanish.
* Patients with severe endometriosis
* Patients with recurrent implantation failure: at least 2 miscarriages or at least 3 transfers with good-quality embryos without pregnancy.
* Patients presenting total fertilization failure or very poor results in any of the two techniques in previous cycles

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Usable blastocyst rate | From oocyte retrieval to 6 days after
  Percentage of oocytes that develop to blastocyst stage and are transferred of cryopreserved
Fertilization rate | From oocyte retrieval to 24 hours later
  Percentage of oocytes that show normal fertilization
Blastocyst rate | From oocyte retrieval to 6 days after
  Percentage of oocytes that develop to blastocyst stage

SECONDARY OUTCOMES:
Pregnancy rate | From embryo transfer to 14 days later
  Percentage of embryo transfers that has a positive beta-hCG 14 days post-transfer
Clinical pregnancy rate | From embryo transfer to 4 weeks later
  Percentage of transfers that have a gestational sac observed 4 weeks post-transfer
Live birth delivery rate | From embryo transfer to 40 weeks later
  Percentage of transfers that end with the delivery of at least one live baby

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico San Carlos, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Who will be able to access the IPD: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
  For what type of analysis: For individual participant data meta-analysis. How they will be able to access: Proposals should be directed to mariadolores.cuquerella@salud.madrid.org. To gain access, data requestors will need to sign a data access agreement.